CLINICAL TRIAL: NCT06851806
Title: A Multicentre, Interventional, Phase IV, Open-label, Study to Evaluate the Safety of Palivizumab in Children Less Than 24 Months of Age With High Risk of Severe Respiratory Syncytial Virus (RSV) Disease
Brief Title: Study of Palivizumab in Children With High Risk of Severe Respiratory Syncytial Virus (RSV) Disease
Acronym: Synagis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: D4800L00014; 2025-000041-13 (EudraCT Number)
Record Dates: First submitted 2025-02-10; First posted 2025-02-28 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Respiratory Syncytial Virus (RSV)
Keywords: Phase IV
MeSH Terms: interventions — Palivizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study Arm (Experimental): All the eligible participants will receive palivizumab 15 mg/kg on Days 1, 31, 61, 91, and 121.
  Interventions: Drug: Palivizumab 15 mg/kg

INTERVENTIONS:
Drug: Palivizumab 15 mg/kg — Single-dose liquid solution vials, 50 mg/0.5 mL, IM injection

SUMMARY:
This is a Phase IV, prospective, open-label, multicentre study to evaluate the safety of palivizumab IM injection for the prevention of severe LRTD in Indian infants and children who are at high-risk of RSV disease. All enrolled participants will receive palivizumab 15 mg/kg IM injection once a month for up to 5 injections during the study. Children who undergo cardiac surgery with cardiopulmonary bypass during the study should receive an additional dose of study intervention immediately after surgery, when medically stable for IM injection as determined by the physician. Prior to each study intervention administration, all participants will undergo safety assessments. A follow-up visit will be performed telephonically with the parent(s) or legal guardian(s) of all participants 30 days after their last injection of palivizumab.

ELIGIBILITY:
Inclusion Criteria:

1. Participants at risk of severe RSV disease defined as fulfilling at least one of the following:

   1. Infants born ≤ 35 wGA and are < 6 months of age at enrolment.
   2. Children < 24 months of age at enrolment and requiring treatment for BPD within the last 6 months.
   3. Children < 24 months of age and with haemodynamically significant CHD.
2. Written informed consent obtained from the participant's parent(s)/legal guardian and the participant's parent(s)/legal guardian is able to understand and comply with the requirements of the protocol including follow-up visits as judged by the investigator.

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

1. Hospitalisation at the time of enrolment, unless the discharge is expected within 30 days of the time of enrolment
2. Required mechanical ventilation (including continuous positive airway pressure) or other mechanical respiratory or cardiac support at the time of enrolment.
3. Anticipated cardiac surgery within 2 weeks after enrolment.
4. Anticipated survival of < 6 months after enrolment in the trial.
5. Active LRTD, including RSV infection at the time of enrolment and/or study intervention administration.
6. Any fever (≥ 38.0°C) or acute illness within 7 days prior to investigational product administration.
7. Known history of evolving or unstable neurologic disorder.
8. Known history of unstable cardiac or respiratory status, including cardiac defects so severe that survival is not expected or for which cardiac transplantation is planned or anticipated.
9. Known allergy, including to immunoglobulin products, or history of allergic reaction.
10. Receipt of palivizumab or other RSV monoclonal antibodies or any RSV vaccine, including maternal RSV vaccination.
11. Receipt of any monoclonal or polyclonal antibody (for example, hepatitis B immune globulin, intravenous immunoglobulin) or anticipated use during the study.
12. Concurrent enrolment in another interventional study.
13. Children of employees of the sponsor, clinical study site, or any other individuals involved with the conduct of the study, or immediate family members of such individuals.
14. Judgment by the investigator that the participant should not participate in the study if the participant or the participant's parent/legal guardian is unlikely to comply with study procedures, restrictions, and requirements.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2025-11-30 (Estimated); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
To assess the safety of palivizumab prophylaxis when administered to preterm infants (≤ 35 wGA), children with BPD (< 24 months) and/or children with haemodynamically significant CHD (< 24 months). | screening to day 151
  1) To determine percentage of participants with AEs and SAEs. 2) To assess nature, incidence, and severity of all AEs including unexpected adverse drug reactions 2)To determine percentage of participants with AEs that lead to study intervention discontinuation.